CLINICAL TRIAL: NCT00980746
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2 093) as Therapy for Patients With Painful Diabetic Neuropathy: a Double-blind, Double-dummy, Randomised, Placebo-controlled, Parallel-group, Multicentre Clinical Trial
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate as Therapy for Patients With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-206; EudraCT 2007-002461-12
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Painful Diabetic Neuropathy
Keywords: pain diabetes neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- ESL 400 mg BID (Experimental): ESL 400 mg twice daily (BID)
  Interventions: Drug: Eslicarbazepine acetate
- ESL 800 mg QD (Experimental): ESL 800 mg once-daily (QD)
  Interventions: Drug: Eslicarbazepine acetate
- ESL 600 mg BID (Experimental): Eslicarbazepine 600 mg twice daily
  Interventions: Drug: Eslicarbazepine acetate
- ESL 1200 mg QD (Experimental): Eslicarbazepine acetate 1200 mg once daily
  Interventions: Drug: Eslicarbazepine acetate
- ESL 800 mg BID (Experimental): Eslicarbazepine acetate 800 mg twice daily
  Interventions: Drug: Eslicarbazepine acetate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine acetate — Eslicarbazepine acetate tablets, scored to allow dose titration during the titration period.
  Other Names: Zebinix
  Arms: ESL 1200 mg QD; ESL 400 mg BID; ESL 600 mg BID; ESL 800 mg BID; ESL 800 mg QD
Drug: Placebo — oral route
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of eslicarbazepine acetate (ESL) as therapy for patients with painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Men and women aged 18 years or older
* Diagnosis of diabetes mellitus Type 1 or 2
* Diagnosis of pain attributed to diabetic neuropathy for more than 1 year prior to enrolment
* Stable glycemic control: (total glycated haemoglobin [HbA1c] level ≤ 11% at screening)
* Cooperation and willingness to complete all aspects of the study
* Completion of at least 4 daily diaries during the week preceding randomisation
* A minimum average daily pain score of 4 on the Numeric rating pain scale (NRPS) in the last 4 diary entries before randomisation.

Exclusion Criteria:

* Pain of other origin that might confound the assessment of neuropathic pain of diabetic origin
* Significant or unstable medical or psychiatric disorders
* Drug or alcohol abuse in the preceding 2 years
* Peripheral vascular disease with a history of amputation, except amputation of toes
* Severe renal function impairment, as shown by calculated creatinine clearance values < 30 mL/min at screening
* Relevant clinical laboratory abnormalities (e.g., Na+ <130 mmol/L, alanine (ALT) or aspartate (AST) transaminases >2.0 times the upper limit of normal, white blood cell count (WBC) <2,500 cells/mm3)
* Previous participation in any study with eslicarbazepine acetate
* Pregnancy or breast feeding
* History of hypersensitivity to the investigational products or to drugs with a similar chemical structure
* History of non-compliance
* Likelihood of requiring treatment during the study period with drugs or other interventions not permitted by the clinical study protocol.
* Participation in a clinical study within 3 months prior to screening
* Any clinically significant concomitant condition, which might influence the assessments or conduct of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date first subject enrolled: 06 Nov 2007 Date last subject completed: 18 Nov 2008 Randomised and treated: 557. Analyzed for efficacy (per-protocol [PP]): 403. Analyzed for safety: 557.
Pre-assignment Details: During the 2week baseline period,current neuropathic pain drug therapy was discontinued and subjects had to be free of any medication that could affect efficacy(except authorized rescue medication)for 2weeks before start of double-blind study treatment.In case of unbearable pain, this drug-free period could be reduced,but had to be at least 7 days.
Groups:
- ESL 1200 mg QD: Eslicarbazepine acetate (ESL) 1200 mg once daily. ESL tablets, scored to allow dose titration during the titration period.
- ESL 400 mg BD: ESL 400 mg twice daily
  ESL tablets, scored to allow dose titration during the titration period.
- ESL 600 mg BID: ESL 600 mg twice daily
  ESL tablets, scored to allow dose titration during the titration period.
- ESL 800 mg BID: ESL 800 mg twice daily
  ESL tablets, scored to allow dose titration during the titration period.
- ESL 800 mg QD: ESL 800 mg once-daily
  ESL tablets, scored to allow dose titration during the titration period.
- Placebo: Placebo
  Placebo : oral route
Period: Overall Study
Arm/Group | ESL 1200 mg QD | ESL 400 mg BD | ESL 600 mg BID | ESL 800 mg BID | ESL 800 mg QD | Placebo
Started | 85 | 89 | 95 | 100 | 92 | 96
Randomized | 85 | 89 | 95 | 100 | 92 | 96
Safety Population | 85 | 89 | 95 | 100 | 92 | 96
Per-protocol | 55 | 66 | 73 | 62 | 73 | 74
Completed | 58 | 67 | 75 | 64 | 75 | 78
Not Completed | 27 | 22 | 20 | 36 | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- ESL 1200 mg QD: Eslicarbazepine acetate 1200 mg once daily
  Eslicarbazepine acetate : Eslicarbazepine acetate tablets, scored to allow dose titration during the titration period.
- ESL 400 mg BD: ESL 400 mg twice daily
  Eslicarbazepine acetate : Eslicarbazepine acetate tablets, scored to allow dose titration during the titration period.
- ESL 600 mg BID: Eslicarbazepine 600 mg twice daily
  Eslicarbazepine acetate : Eslicarbazepine acetate tablets, scored to allow dose titration during the titration period.
- ESL 800 mg BID: Eslicarbazepine acetate 800 mg twice daily
  Eslicarbazepine acetate : Eslicarbazepine acetate tablets, scored to allow dose titration during the titration period.
- ESL 800 mg QD: ESL 800 mg once-daily
  Eslicarbazepine acetate : Eslicarbazepine acetate tablets, scored to allow dose titration during the titration period.
- Total: Total of all reporting groups
Arm/Group | ESL 1200 mg QD | ESL 400 mg BD | ESL 600 mg BID | ESL 800 mg BID | ESL 800 mg QD | Placebo | Total
Number analyzed (Participants) | 85 | 89 | 95 | 100 | 92 | 96 | 557
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 61 | 61 | 61 | 59 | 65 | 360
  >=65 years | 32 | 28 | 34 | 39 | 33 | 31 | 197
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 56 | 56 | 50 | 57 | 309
  Male | 43 | 41 | 39 | 44 | 42 | 39 | 248

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Mean Pain, Scored Daily on a on an 11-point (0-10) Numeric Rating Pain Scale (NRPS), Where 0 = no Pain and 10 = Worst Possible Pain
Description: Endpoint mean pain was defined as the mean of the last 4 available pain scores in the last 7 days of the treatment period. Likewise, baseline mean pain was defined as the mean of the last 4 available pain scores in the last 7 days of the baseline period.
Time Frame: 17 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ESL 1200 mg QD | ESL 400 mg BD | ESL 600 mg BID | ESL 800 mg BID | ESL 800 mg QD | Placebo
Number analyzed (Participants) | 85 | 89 | 95 | 100 | 92 | 96
units on a scale | -1.7546 (0.2352) | -2.2865 (0.2325) | -1.6746 (0.2312) | -1.8353 (0.2260) | -1.9829 (0.2328) | -1.5801 (0.2311)

ADVERSE EVENTS:
Time Frame: All Treatment-emergent adverse event (TEAEs), i.e. those Adverse events (AEs) starting after the first dose intake until 2 days after the last dose,have been summarized
Arm/Group | ESL 1200 mg QD | ESL 400 mg BD | ESL 600 mg BID | ESL 800 mg BID | ESL 800 mg QD | Placebo
Serious Adverse Events (participants affected / at risk) | 7/85 | 3/89 | 0/95 | 4/100 | 1/92 | 0/96
Other Adverse Events (participants affected / at risk) | 11/85 | 0/89 | 23/95 | 35/100 | 0/92 | 6/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESL 1200 mg QD (N=85) | ESL 400 mg BD (N=89) | ESL 600 mg BID (N=95) | ESL 800 mg BID (N=100) | ESL 800 mg QD (N=92) | Placebo (N=96)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESL 1200 mg QD (N=85) | ESL 400 mg BD (N=89) | ESL 600 mg BID (N=95) | ESL 800 mg BID (N=100) | ESL 800 mg QD (N=92) | Placebo (N=96)
Nausea (General disorders) | 0 (0) | 0 (0) | 7 (7) | 10 (10) | 0 (0) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 0 (0) | 5 (5) | 9 (9) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other